CLINICAL TRIAL: NCT02225977
Title: Assessing Induction of Type II (M2) Monocytes/Macrophages in Patients Receiving Gilenya.
Status: Completed | Type: Observational
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Brett T. Lund, Assistant Professor of Neurology, University of Southern California
Other Study IDs: MSGilenya
Record Dates: First submitted 2014-08-24; First posted 2014-08-26 (Estimated); Last update posted 2018-08-22 (Actual); Status verified 2018-08

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Fingolimod Hydrochloride

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- Gilenya treated - 1 month: Patient's taking continuous oral Gilenya at prescribed dose for 1 month.
  Interventions: Drug: Gilenya
- Gilenya treated - 3 months: Patient's taking continuous oral Gilenya at prescribed dose for 3 months.
  Interventions: Drug: Gilenya
- Gilenya treated - 6 months: Patient's taking continuous oral Gilenya at prescribed dose for 6 months.
  Interventions: Drug: Gilenya
- Gilenya treated - 12 months: Patient's taking continuous oral Gilenya at prescribed dose for 12 months.
  Interventions: Drug: Gilenya
- Gilenya qualified - untreated: Patient's qualifying to start treatment with oral Gilenya at prescribed dose but still as yet untreated.

INTERVENTIONS:
Drug: Gilenya
  Groups: Gilenya treated - 1 month; Gilenya treated - 12 months; Gilenya treated - 3 months; Gilenya treated - 6 months

SUMMARY:
In this study we wish to test the hypothesis that continuous Gilenya treatment alters immune homeostasis in favor of an anti-inflammatory type II monocyte and macrophage (M2) phenotype in the circulation of patients with relapsing-remitting Multiple Sclerosis (MS). In this study we will determine the change in ratio of M2 (type II, alternatively activated) versus M1 (type I, classically activated) monocytes and macrophages in a cohort of patients that have received continuous Gilenya treatment for 0, 1, 3, 6 or 12 months. We will also assess changes in cell surface expression of the M1 marker CCR7 and the M2 markers CD206 or CD301 by monocytes and macrophages using FACS analysis of whole blood, and assess the tyrosine phosphorylation of the signal transducer and activator of transcription STAT-1 (pTyr-STAT1), which is critical for the activation of M1 myeloid cells. We will assess correlates with changes in M1 and M2 cytokine expression assessing possible mechanisms of action of Gilenya on myeloid lineage cells.

ELIGIBILITY:
Inclusion Criteria:

* Patients must qualify to receive treatment with Gilenya, according to the University of Southern California, Department of Neurology, MS Group, Gilenya Prescribing Process.
* Clinically definite Multiple Sclerosis defined by the revised McDonald criteria (Polman et al., 2005, Polman et al., 2010) of the relapsing-remitting form with an Expanded Disability Status Scale (EDSS) score of 0 to 5.5.
* Ability to understand and sign this study-specific institutional review board-approved informed consent form.
* Willing to donate ~50mls of blood for immunological testing on up to five occasions.

Exclusion Criteria:

* Patient does not qualify to receive treatment with Gilenya, according to the USC, Department of Neurology, MS Group, Gilenya Prescribing Process.
* Inability to understand nature of the study.
* Treatment with any of the following within 30 days of commencing treatment with Gilenya: Avonex, Betaseron, Rebif, Copaxone, Natalizumab, Rituximab, Mitoxantrone, Cyclophosphamide, Cyclosporine, Azathioprine, Methotrexate or any other immunomodulatory, immunosuppressant or immune homeostasis altering drug.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be selected from those seen by physicians at the USC Multiple Sclerosis Comprehensive Care Center.
Sampling Method: Non-Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2013-07-31 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2017-04-30 (Actual)

PRIMARY OUTCOMES:
Change in ratio of M2 versus M1 monocytes and macrophages. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Brett T Lund, Ph.D., Principal Investigator — University of Southern California
Locations (1):
- University of Southern California, Department of Neurology, Los Angeles, California, United States